CLINICAL TRIAL: NCT03745092
Title: The Efficacy of Normobaric Oxygen on Chronic Cerebral Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ran Meng, Principal investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NBO-CCI
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Normobaric Oxygen; Cerebral Ischemia
Keywords: normobaric oxygen; cerebral ischemia; EEG
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO group (Experimental): Between the two time 30min-EEG recordings, the patients in the NBO group would receive NBO (8L/min, via face mask) for 45min.
  Interventions: Device: normobaric oxygen
- Control group (Placebo Comparator): Between the two time 30min-EEG recordings, the patients in the control group would have a rest (lying, sitting or walking) for 45min.
  Interventions: Device: room air

INTERVENTIONS:
Device: normobaric oxygen — Normobaric oxygen (NBO) is a routine adjuvant hyperoxygenation intervention supplied by facemask (such as Venturi mask), with one atmosphere pressure (1ATA=101.325kPa).
  Arms: NBO group
Device: room air — The patient had a rest with lying, sitting or walking, did not performed with NBO intervention.
  Arms: Control group

SUMMARY:
Chronic cerebral ischemia (CCI) is viewed as an alarming state induced by long-term reduction in cerebral perfusion, which is associated with neurological deficits and high risk of stroke occurrence or recurrence. CCI accounts for a large proportion in both outpatient and inpatient subjects with cerebrovascular disease, while the treatment of CCI remains a formidable challenge to clinicians. Normobaric oxygen (NBO) is an adjuvant hyper-oxygenation intervention supplied with one atmosphere pressure (1ATA=101.325kPa). A plethora of studies have demonstrated the efficacy of NBO on the penumbra in acute stroke. NBO has been shown to increase oxygen pressure, raise intracranial blood flow, protect blood-brain barrier and enhance neuro-protective effects. As the similar underlying mechanisms shared by the penumbra in stroke and the ischemic-hypoxic brain tissues in CCI, the investigators speculate that NBO may serve as a promising therapeutic strategy for attenuating short-term symptoms or improving long-term clinical outcomes amongst patients with CCI. Due to the scant research exploring the efficacy of NBO for treating CCI so far, the clinical studies are warranted to verify this hypothesis urgently.

DETAILED DESCRIPTION:
INTRODUCTION Chronic cerebral ischemia (CCI), which is firstly proposed by Japanese scholars in 1990s, is considered as a pathological status induced by persistent reduction of cerebral blood volume and flow (CBV and CBF), leading to ischemia and hypoxia in the brain tissue. Long-time ischemic-hypoxic injury can cause various atypical brain dysfunctions, such as headache, dizziness, cognitive decline and emotional abnormalities. Under the low-perfusion background, the brain tissue is more vulnerable to ischemic-hypoxic insult; thus, the incidence of ischemic events amongst individuals with CCI is substantially higher than those without. It has been reported that intracranial atherosclerotic stenosis (ICAS), internal jugular venous stenosis (IJVS) and cardiogenic cerebral circulation insufficiency are the common pathogenesis of CCI, with the hypoperfusion as a vital mechanism accounting for these clinical presentations.

Normobaric oxygen (NBO) is a routine adjuvant hyperoxygenation intervention supplied by nasal cannula or facemask (such as Venturi mask), with one atmosphere pressure (1ATA=101.325kPa). Evidence available shows that NBO may be a safe, convenient and promising therapeutic strategy for multi-organ protection, which has garnered increasing attention of researchers over the past years. However, some studies do not support the favorite efficacy of NBO. For instance, a large meta-analysis conducted by Chu et al. revealed that in acutely ill adult patients, oxygen supplementation might increase mortality without improving patient-important outcomes. The negative results can contribute to acute critical conditions and some serious complications such as infection, arrhythmia and dyspnea. In contrast to previous experimental data confirming the NBO protection on acute stroke, a recent multi-center randomized clinical trial concludes that this oxygen supplement does not reduce the rate of death or disability. The incongruent conclusions between clinical and animal studies may be attributable to the protective mechanisms of NBO behind cerebral ischemia, the rationale for the protective effect afforded by NBO is freezing penumbra and extending the time window for reperfusion, meaning that NBO may be not applicable for patients with permanent vessel occlusion. Animal research has corroborated that NBO can reduce infarct size and improve post-stroke outcomes after thrombolysis in ischemic stroke, and a large multi-center randomized prospective trial is ongoing.

Theoretically, low cerebral blood perfusion in CCI patients exposes the brain tissue to an ischemic-hypoxic condition, which is similar to that in penumbra in acute ischemic stroke. Therefore, given the prominent effectiveness in penumbra, NBO, which can supply abundant oxygen, may yield some benefits to the ischemic-hypoxic brain tissue in CCI patients. However, there is no study investigating the oxygen supplementation applied in CCI up to now.

THEORY OF THE HYPOTHESIS

The investigators' hypothesis is that NBO can enhance oxygen content in the ischemic-hypoxic brain tissue in CCI patients and subsequently improve both short-term symptoms and long-term clinical outcomes. The basis of the hypothesis is inferred by several convinced theories presented as follows:

1. NBO is capable of increasing the arterial partial pressure of oxygen (pO2) and raising the dissolved oxygen fraction in the aorta and the smallest arterioles. In this regard, Liu et al. reported that after NBO treatment, the penumbral interstitial pO2 could be maintained close to pre-ischemic normal value. Given the fact that both penumbra in acute stroke and abnormal brain tissues in CCI are caused by ischemia and hypoxia, NBO may be conceived as an effective adjuvant therapy for CCI as well.
2. NBO can increase CBF/CBV in the penumbra in acute stroke. During NBO treatment, vasodilation occurs in the ischemic regions, while the non-ischemic regions show vasoconstriction. The raised pO2 and increased blood flow in the penumbra are involved in down regulating zinc levels, which may contribute to the neuro-protective effect by NBO. Whereby, improving perfusion in the ischemic-hypoxic brain tissue can result in the relief of the associated clinical symptoms.
3. NBO is able to attenuate blood brain barrier (BBB) disruption in cerebral ischemia, possibly through inhibiting matrix metalloproteinase-9 (MMP-9) mediated degradation of tight junction proteins. The integrity of BBB is influenced by various pathological processes, such as inflammatory mediators invasion, edema formation, and hemorrhagic transformation. Similarly, BBB protection provided by NBO may also be available to CCI patients so that the impaired brain functions may be at least partially restored, or delayed CCI-induced brain damage.
4. Other underlying neuro-protective mechanisms, including reducing peri-infarct depolarizations, improving aerobic metabolism, preventing apoptotic cell death and ameliorating inflammation can offer benefits to patients with cerebral ischemia. On the other hand, NBO is safe enough as it does not augment the formation of reactive oxygen species, nitrogen species and some other mediators implicated in the exacerbation of oxidative stress injury.

Currently, there are very few reports in literature regarding the application of NBO in CCI and this is undoubtedly a brand-new field that deserves more attention. Differ from the beneficial effects observed in experimental stroke models, most of the clinical trials failed to reach favorable results. As the investigator discussed aforementioned, the ischemic penumbra is a vital target for NBO and low rate of revascularization is responsible for the poor outcomes in acute stroke patients. CCI refers to a state of long-term reduction in cerebral perfusion secondary to ICAS, IJVS or other pathogeneses, meaning that most of the afflicted brain tissues are in ischemic-hypoxic conditions, just like the penumbra in acute stroke. This phenomenon suggests that supplying enough oxygen may hold the potential of enhancing the resistance of brain tissues to hypoxic insults, slowing down the deterioration and preventing secondary ischemic stroke in CCI patients. Meanwhile, rapid oxygen content enhancement enables immediate improvements in ischemic-hypoxic conditions, allowing for the relief of clinical symptoms in a short period of time.

IMPLICATIONS OF THE HYPOTHESIS In real clinical practice, there are a large number of patients suffering from CCI and the current mainstay therapeutic strategies are far from satisfactory. Conservative therapies mainly involve anti-platelets, lipid-lowering agents and neuro-protectives, but their effectiveness is still uncertain. The efficacy of endovascular treatment, such as endarterectomy and intravascular stenting, is still controversial and should not be considered superior to the conservative treatment. Moreover, endovascular treatment may be not suitable for all patients with CCI. Recently, remote ischemic conditioning (RIC) has emerged as an innovative and promising adjunctive approach for multi-organ protection. It has been demonstrated that daily RIC can reduce the rate of stroke recurrence and improve the long-term clinical outcomes in patients with CCI. However, it is reasonable to expect that RIC requires a longer time to take effect, thus patients cannot relieve their symptoms within a short period of time following treatment initiation. Meanwhile, there is still a portion of patients who may not benefit from or be contraindicated to RIC. According to available evidence and the hypothesis, NBO is able to enhance the oxygen content of ischemic regions, increase cerebral perfusion, and prevent brain tissues from secondary injury, all of which could help relieve the symptoms in a short time and improve the long-term clinical outcomes profoundly. Therefore, NBO may serve as a promising adjunctive alternative to current treatment strategies.

CONCLUSION As NBO may profoundly improve both the short-term symptoms as well as the long-term clinical outcomes in CCI patients, it should be deemed as a brand-new effective and convenient adjuvant treatment strategy if the hypothesis is validated. Well-designed animal experiments and clinical trials are urgently warranted in the next step to corroborate the effectiveness of NBO on brain protection in patients with CCI.

ELIGIBILITY:
Inclusion criteria: (1) age from 18 to 80 years; (2) diagnosis of intracranial arterial stenosis or internal carotid arterial stenosis; (3) NIHSS≤4 and mRS≤2; (4) signed informed consent.

Exclusion criteria: (1) brain infarction occurring within recent two months; (2) intracranial arterial aneurysm, dissection or malformation; (3) history of cerebral hemorrhage or subarachnoid hemorrhage; (4) history of cerebral trauma; (5) history of other brain injury or disorders; (6) austere diseases such as cancer, heart failure, respiratory failures; (7) respiratory diseases; (8) poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Captial Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
including the number of enrolled cases, the primary outcomes and the second outcomes.
Supporting Information: SAP, CSR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NBO Group | Control Group
Started | 26 | 23
Completed | 26 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NBO Group | Control Group | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 38
  >=65 years | 9 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (8.3) | 55.0 (8.4) | 56.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 18 | 19 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 26 | 23 | 86

OUTCOME MEASURES:

1. Primary Outcome: The Fronto-central Theta Absolute Power Change Rate
Description: The patients undergo 30-minute EEG recordings two times. Between the two times of EEG recordings, the patients are performed with the specific interventions (NBO or rest) for 45 minutes. The fronto-central theta absolute power change rate was calculated as the theta (4-8Hz) absolute power at (the baseline EEG minus the post-intervention EEG)/the baseline EEG over the fronto-central electrodes (F3, F4, Fz, C3, C4, Cz). The theta absolute power (with units microvolts squared) is computed using Fast Fourier Transform for each electrode over the theta frequency band.
Time Frame: 30 minutes baseline EEG, 45 minutes intervention, 30 minutes post-intervention EEG
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 26 | 23
ratio | 0.14 [-0.07 to 0.37] | -0.12 [-0.24 to 0.04]

2. Primary Outcome: The Fronto-central Delta Absolute Power Reduction Rate
Description: The patients undergo 30-minute EEG recordings two times. Between the two times of EEG recordings, the patients are performed with the specific interventions (NBO or rest) for 45 minutes. The fronto-central delta absolute power change rate was calculated as the delta (1-4Hz) absolute power at (the baseline EEG minus the post-intervention EEG)/the baseline EEG over the fronto-central electrodes (F3, F4, Fz, C3, C4, Cz). The delta absolute power (with units microvolts squared) is computed using Fast Fourier Transform for each electrode over the delta frequency band.
Time Frame: 30 minutes baseline EEG, 45 minutes intervention, 30 minutes post-intervention EEG
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 26 | 23
ratio | 0.21 [0.07 to 0.38] | -0.01 [-0.20 to 0.15]

3. Secondary Outcome: The Post-intervention Fronto-central Theta/Alpha Ratio
Description: The patients undergo 30-minute EEG recordings two times. Between the two times of EEG recordings, the patients are performed with the specific interventions (NBO or rest) for 45 minutes. The post-intervention fronto-central theta/alpha ratio is computed as the theta absolute power/the alpha absolute power over the fronto-central electrodes (C3, C4, Cz, F3, F4, Fz) at the post-intervention EEG. The alpha and theta absolute power (with units microvolts squared) is computed using Fast Fourier Transform for each electrode over the alpha (8-12Hz) and theta (4-8Hz) frequency band.
Time Frame: 30 minutes baseline EEG, 45 minutes intervention, 30 minutes post-intervention EEG
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 26 | 23
ratio | 0.36 [0.16 to 0.49] | 0.35 [0.21 to 0.79]

4. Secondary Outcome: The Post-intervention Fronto-central (Delta+Theta)/(Alpha+Beta) Ratio
Description: The patients undergo 30-minute EEG recordings two times. Between the two times of EEG recordings, the patients are performed with the specific interventions (NBO or rest) for 45 minutes. The post-intervention fronto-central (delta+theta)/(alpha+beta) ratio is computed as (the delta+theta absolute power)/(the alpha+beta absolute power) over the fronto-central electrodes (C3, C4, Cz, F3, F4, Fz) at the post-intervention EEG. The beta, alpha, theta and delta absolute power (with units microvolts squared) is computed using Fast Fourier Transform for each electrode over the beta (12-20Hz), alpha (8-12Hz), theta (4-8Hz) and delta (1-4Hz) frequency band.
Time Frame: 30 minutes baseline EEG, 45 minutes intervention, 30 minutes post-intervention EEG
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 26 | 23
ratio | 0.64 [0.34 to 0.92] | 0.58 [0.42 to 1.29]

5. Secondary Outcome: The Post-intervention Fronto-central Delta/Alpha Ratio
Description: The patients undergo 30-minute EEG recordings two times. Between the two times of EEG recordings, the patients are performed with the specific interventions (NBO or rest) for 45 minutes. The post-intervention fronto-central delta/alpha ratio is computed as the delta absolute power/the alpha absolute power over the fronto-central electrodes (C3, C4, Cz, F3, F4, Fz) at the post-intervention EEG. The alpha and delta (1-4Hz) absolute power (with units microvolts squared) is computed using Fast Fourier Transform for each electrode over the alpha (8-12Hz) and delta (1-4Hz) frequency band.
Time Frame: 30 minutes baseline EEG, 45 minutes intervention, 30 minutes post-intervention EEG
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 26 | 23
ratio | 0.33 [0.18 to 0.80] | 0.35 [0.29 to 0.62]

6. Secondary Outcome: The Fronto-central Wavelet Entropy Change
Description: The entropy is computed via nonlinear dynamics method and represents the complexity of the signal in the information science initially (with units nat). It can also be applied in assessing the complexity of the EEG signal to evaluate the brain functions. The wavelet entropy analysis is a sub-type of entropy which is proceeded with wavelet transform. The wavelet entropy analysis provides a quantitative measure of the degree of disorder in the brain rhythm at various times in brain injury and recovery. The higher value of the wavelet entropy indicates the better brain functions. The fronto-central wavelet entropy change in this study is defined as the wavelet entropy value at the baseline EEG minus the post-intervention EEG over the fronto-central electrodes (F3, F4, Fz, C3, C4, Cz).
Time Frame: 30 minutes baseline EEG, 45 minutes intervention, 30 minutes post-intervention EEG
Measure: Mean (Standard Deviation); unit: nat
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 26 | 23
nat | -0.15 (0.54) | -0.01 (0.42)

ADVERSE EVENTS:
Time Frame: 4 months
Description: All of the participants were with NIHSS≤4 and mRS≤2. NBO was supplied with 8L/min for 45min between the two times EEG recordings. Short-term performance, low flow velocity and mild neurological disorders rendered our intervention enough safe for the participants. All of the participants were followed up for 4 months and seven of them were performed with NBO with 5L/min, 45 minutes each time, 3 times daily, they did not reported any adverse events.
Arm/Group | NBO Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03745092/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03745092/ICF_001.pdf